CLINICAL TRIAL: NCT00841620
Title: Symptom Control 1-year After Circular Stapler Anopey or Diathermy Excision for Prolapsed Haemorrhoids: an International Randomsed Trial (the STOPP-trial
Brief Title: Symptom Control 1-year After Circular Stapler Anopexy or Diathermy Excision for Prolapsed Haemorhoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Niels Qvist, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOPP
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Hemorrhoids
Keywords: Symptoms; Postoperative pain; Postoperative complications; Milligan; Anopxy
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Haemorrhoidectomy a.m. Milligan for grade 3-4 haemorrhoids
  Interventions: Procedure: Haemorrhoidectomy a.m. Milligan
- 2 (Active Comparator): Stapled anopexy for grade 3-4 haemorrhoids
  Interventions: Procedure: Stapled anopexy

INTERVENTIONS:
Procedure: Haemorrhoidectomy a.m. Milligan — Surgery
  Arms: 1
Procedure: Stapled anopexy — Surgery
  Arms: 2

SUMMARY:
Background: In an international randomised controlled trial we studied how patient self-reported symptoms improved after either a stapled anopexy operation or a diathermy excision of the haemorrhoids.

Methods: The study involved 18 hospitals in Sweden, Denmark and the UK. Two hundred and seven patients were randomised. After exclusion of 27 patients, 90 in both groups were operated and followed one year. Patients provided self-reported symptoms before surgery and after 1 year. A patient diary obtained daily self-reported postoperative pain scores (VAS). Surgeons evaluated the anal anatomy before surgery and after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Grades III and IV haemorrhoids

Exclusion Criteria:

* Previous operation for high anal fistula or injury to the anal sphincteres

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 1999-09; Primary Completion 2001-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Self-reported frequency of symptoms | one year

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Principal Investigator
Locations (1):
- Odense University Hospital, Odense C, Denmark